CLINICAL TRIAL: NCT05576038
Title: Restoration of Impaired Microbiota-mediated Aryl Hydrocarbon Receptor Signaling in Celiac Disease by Oral Tryptophan Supplementation: an Exploratory, Pilot Trial
Brief Title: Tryptophan for Impaired AhR Signaling in Celiac Disease
Acronym: TIARSCeD
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: McMaster University (Other)
Responsible Party: Principal Investigator, David Armstrong, Professor of Medicine, McMaster University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 14582
Record Dates: First submitted 2022-10-03; First posted 2022-10-12 (Actual); Last update posted 2025-01-10 (Actual); Status verified 2025-01

CONDITIONS: Tryptophan Metabolism Alterations; Celiac Disease
Keywords: Tryptophan; Celiac disease; Aryl Hydrocarbon Receptor
MeSH Terms: conditions — Celiac Disease | interventions — Tryptophan

STUDY DESIGN:
Intervention Model Description: Prospective randomized controlled trial: double-blinded, placebo controlled exploratory study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Interventions will be blinded by McMaster University Central Pharmacy
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- L-Tryptophan (Active Comparator): L-tryptophan* supplements (Tryptan, Valeant Canada LP): each treatment capsule contains 500 mg of L-Tryptophan; talc and magnesium stearate.
  Study participants will be instructed to take 2 x 500 mg capsules (1000 mg) every 8 hrs, three times a day. (total daily dose: 3000 mg) for a total of 3 weeks.
  Instructions will be printed on the label of the pill container.
  Interventions: Drug: L-Tryptophan
- Freedom SimpleCap Powder (Placebo Comparator): 500 mg of SimpleCap Powder. Study participants will be instructed to take 2 x 500 mg capsules (1000 mg) every 8 hrs, three times a day. (total daily dose: 3000 mg) for a total of 3 weeks.
  Instructions will be printed on the label of the pill container.
  Interventions: Drug: Freedom SimpleCap Powder

INTERVENTIONS:
Drug: L-Tryptophan — L-tryptophan is an essential amino acid responsible for activating the aryl hydrocarbon receptor (AhR). Dietary tryptophan is metabolized by the gut microbiota producing several 'indoles' such as (indole-3-aldehyde (IAld), indole-3-acetic acid (IAA), indole-3 propionic acid (IPA), indole-3-acetaldehyde (IAAld), indole-3-lactic acid (ILA) and indole-acrylic acid) and tryptamine, which are ligands for the AhR, a nuclear transcription factor involved in activating target genes responsible for maintaining gut integrity. Prior literature suggests that patients with active celiac disease have a lower functional capacity to produce these AhR ligands, which further impairs the AhR pathway. Hence, the aim of this study is to assess the effects of tryptophan supplementation in patients with celiac disease, non-responsive to a GFD for more than 1 year compared with the effects of an inactive, placebo comparator, L-leucine.
  Arms: L-Tryptophan
Drug: Freedom SimpleCap Powder — Freedom SimpleCap Powder is a high functionality capsule and tablet excipient composite comprised of filler, glidant, disintegrant and lubricant (ingredients include: Microcrystalline Cellulose, Silicon Dioxide Colloidal, Sodium Starch Glycolate, Sodium Stearyl Fumarate). This capsule is dye, lactose and gluten free and will not interfere with the AhR pathway. Freedom SimpleCap Powder makes oral capsule formulation convenient, quick and simple Thus, this SimpleCap Powder will be an appropriate placebo comparator for this study.
  Arms: Freedom SimpleCap Powder

SUMMARY:
This is a prospective, randomized, double-blind, placebo-controlled exploratory trial to evaluate the effect of L-tryptophan supplementation on celiac-related symptoms in individuals who have biopsy-confirmed celiac disease (CeD) and symptoms non-responsive to a gluten-free diet (GFD). Fifty participants, aged 18 to 75 years, who self-report persistent CeD-related symptoms despite taking a GFD for more than 1 year and who score > 40 on the Celiac Symptom Index (CSI) will be randomized to receive L-tryptophan or placebo for 3 weeks.

DETAILED DESCRIPTION:
At Visit 1, consented participants will receive study instructions and be randomized 1:1 to L-tryptophan or placebo (SimpleCap). A dietitian will counsel all 50 participants on how to maintain a low tryptophan, gluten-free diet. This diet provides an adequate intake of protein (50 g/day) and energy (1800 kcal/day) while limiting the consumption of high tryptophan-containing foods. Study participants will receive all their intervention capsules at Visit 1 to be taken for 3 weeks, starting the day after Visit 2. At Visits 2 and 3, just before and after the intervention, participants will complete dietary and symptom questionnaires, provide blood, stool, and urine samples, and undergo upper endoscopy to obtain aspirates from the second part of the duodenum, using a sterile catheter followed by six duodenal biopsies, 2 from the first part (bulb) and 4 from the second part of the duodenum. Dietary compliance will be assessed 3-day recalls which will further be analysed by using ESHA Food Processor, a Nutritional Analysis Software.

ELIGIBILITY:
Inclusion criteria:

* 18 and 75 years of age
* Celiac disease (CeD) diagnosis: Individuals with histological and serological evidence of CeD serology (positive biopsy and anti-tTG IgA)
* Persistent CeD related symptoms (>40 on the Celiac Symptom Index) despite >1 year of a gluten free diet (GFD)

Exclusion criteria:

* Acid anti-secretory and antacid medications
* Antibiotics, antibacterial agents or probiotics, currently, or within the last 8 weeks
* Current organic gastrointestinal or other autoimmune diseases, such as inflammatory bowel disease or diabetes mellitus (type 1)
* Lactose and/or fructose intolerance
* History of bariatric surgery, fundoplication or gastrectomy (partial or complete)
* Connective tissue disease
* Concurrent organic GI pathology other than benign polyps, haemorrhoids, lipomas, Helicobacter pylori infection, diverticulosis and melanosis coli
* Chronic treatment with high dose opioids
* Alcohol or drug abuse
* Concurrent systemic disease and/or laboratory abnormalities considered by investigators to be a risk or that could interfere with data collection
* Allergy or sensitivity to any component of the study medication or placebo
* Use of lithium and monoamine oxidase inhibitors (MAOIs)
* Participation in another dietary treatment study within the last 4 weeks

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2025-04-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of Celiac Symptom Index (CSI) | 3 weeks
  Change in CSI score; a 7-point decrease in CSI score indicates meaningful improvement.

SECONDARY OUTCOMES:
Patient Assessment of Upper Gastrointestinal Disorders-Quality of Life questionnaire (PAGI-QoL). | 3 weeks
  Change in PAGI-QoL score from baseline to week 3; an increase in score indicates an improvement in quality of life. PAGI-QoL score ranges from 0 to 5, 0 being the lowest and 5 being the highest.
Hospital Anxiety and Depression Scale (HADS) | 3 weeks
  Change in the anxiety and depression scores for the HADS from baseline to week 3; a decrease in the scores indicate decreases in anxiety and depression respectively. The anxiety and depression scales score separately, each ranging from 0 to 21, 0 being the lowest and 21 being the highest.
Gastrointestinal Symptoms Rating Scale (GSRS) | 3 weeks
  Change in GSRS score from baseline to week 3. Score ranges from 1-7; decrease in score indicates improvement.
Intestinal indole production in the duodenum | 3 weeks
  Change in duodenal indole production from baseline to week 3

OTHER OUTCOMES:
Duodenal mucosal villus-crypt ratio (VCR) | 3 weeks
  Change in the duodenal mucosal VCR from baseline to week 3; an increase in the mucosal VCR ratio indicates decreased mucosal injury
Aryl hydrocarbon Receptor (AhR) activation in the duodenum | 3 weeks
  Change in duodenal mucosal AhR activation from baseline to week 3
Tissue transglutaminase IgA (tTG) titres | 3 weeks
  Change in tTG titers from baseline to week 3; a decrease in tTG titres is associated with decreased gluten exposure and, hence, with decreased celiac disease activity

CONTACTS AND LOCATIONS:
Locations (1):
- McMaster University, Hamilton, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No
Data will not be shared among other researchers.